CLINICAL TRIAL: NCT00263718
Title: Calcipotriol Plus Betamethasone Dipropionate Gel Compared to Betamethasone Dipropionate in the Gel Vehicle, Calcipotriol in the Gel Vehicle and the Gel Vehicle Alone in Psoriasis Vulgaris
Brief Title: Efficacy and Safety of Calcipotriol Plus Betamethasone Dipropionate Gel in Psoriasis Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MBL 0202 INT
Record Dates: First submitted 2005-12-08; First posted 2005-12-09 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2015-03

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — calcipotriene; betamethasone-17,21-dipropionate; Gels

INTERVENTIONS:
Drug: Calcipotriol plus betamethasone dipropionate (LEO 80185) gel

SUMMARY:
The objective of the study is to compare the use of calcipotriol plus betamethasone dipropionate gel with betamethasone dipropionate in the gel vehicle, calcipotriol in the gel vehicle and the gel vehicle alone when used in patients with psoriasis vulgaris on the trunk and/or limbs. Patients will be treated once daily for up to 8 weeks.

The primary response criterion is the number of patients with controlled disease at week 8.

ELIGIBILITY:
Inclusion Criteria:

* Psoriasis vulgaris involving trunk and/or arms and/or legs amenable to treatment with a maximum of 100 g of topical medication per week
* An investigators' global assessment of disease severity of at least mild

Exclusion Criteria:

* PUVA or Grenz ray therapy within 4 weeks prior to randomisation
* UVB therapy within 2 weeks prior to randomisation
* Systemic treatment with biological therapies, with a possible effect on psoriasis vulgaris within 6 months prior to randomisation
* Systemic treatment with all other therapies than biologicals, with a possible effect on psoriasis vulgaris (e.g., corticosteroids, vitamin D analogues, retinoids, immunosuppressants) within 4 weeks prior to randomisation
* Any topical treatment of the trunk/limbs (except for emollients) within 2 weeks prior to randomisation
* Topical treatment for other relevant skin disorders (except WHO group I-II corticosteroids, tar, retinoid and dithranol on face, scalp, or flexures) within 2 weeks prior to randomisation
* Planned initiation of, or changes to concomitant medication that could affect psoriasis vulgaris (e.g., beta blockers, anti-malaria drugs, lithium) during the study
* Current diagnosis of guttate, erythrodermic, exfoliative or pustular psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360
Dates: Start 2005-12; Study Completion 2006-05

PRIMARY OUTCOMES:
Patients with "controlled disease" (minimal or clear and at least two steps change from baseline) according to the investigators' global assessment of disease severity at week 4 and week 8.

SECONDARY OUTCOMES:
The absolute and percentage change in PASI from baseline to week 1, 2, 4, 6, and 8.
Patients with "controlled disease" according to the investigators' global assessment of disease severity at week 1, 2, and 6.
Patients with "clear" or "very mild" disease by the patient's global assessment of disease severity at week 1, 2, 4, 6, and 8.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Fleming, MD, Principal Investigator — Ninewells Hospital and Medical School, Ninewells, Dundee, UK
Locations (5):
- The Guenther Dermatology Research Centre, London, Ontario, Canada
- Universitätsklinikum Leipzig, Leipzig, Germany
- Waterford Regional Hospital, Waterford, Ireland
- Läkarhuset Vällingby, Vällingby, Sweden
- Ninewells Hospital and Medical School, Dundee, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en